CLINICAL TRIAL: NCT03416140
Title: Effectiveness and Safety of the Therapeutic Exercise in Patients With Chronic Kidney Disease
Brief Title: Effectiveness Chronic Kidney Disease & Therapeutic Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, PhD, MSc, PT, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERC_ULE_II
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Kidney Diseases; Exercise
MeSH Terms: conditions — Kidney Diseases; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise (Experimental)
  Interventions: Other: Therapeutic Exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Therapeutic Exercise — 30 minutes per day of therapeutic exercise
  Arms: Therapeutic exercise

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of the therapeutic exercise effects in patients with chronic kidney disease. An randomized clinical trial is carried out. A total sample of 70 patients with chronic kidney disease is recruited and divided into a therapeutic exercise group and a control group. The kidney function (creatinine clearance as main outcome) is measured at baseline and 1 month after treatment start.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease

Exclusion Criteria:

* Cognitive impairment and non signed consent inform form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Kidney function | Change from Baseline creatinine clearance at 1 month
  Creatinine clearance

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Neyra Bohórquez, MD, Principal Investigator — Nephrology Unit, Galdakao Hospital, Spain
Locations (1):
- Pierre Neyra Bohórquez, Galdakao, Bizkaia, Spain